CLINICAL TRIAL: NCT04317729
Title: Evaluation of Hepatitis C Virus Antibody Detection From Dried Blood Spots With the Fujirebio INNOTEST® HCV Ab IV
Brief Title: DBS Evaluation of Fujirebio INNOTEST® HCV Ab IV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HC016
Record Dates: First submitted 2019-12-19; First posted 2020-03-23 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (Experimental): Collection of whole blood via fingerstick and venipuncture
  Interventions: Device: Fujirebio INNOTEST® HCV Ab IV assay

INTERVENTIONS:
Device: Fujirebio INNOTEST® HCV Ab IV assay — Enzyme Immunoassay

SUMMARY:
The goal of this trial is to evaluate the performance of the Fujirebio INNOTEST® HCV Ab IV using simpler collection methods such as fingerstick and venous whole blood collection on dried blood spots (DBS). In order to assess performance in samples with high and low antibody titres, performance will be evaluated with undiluted samples of all trial participants and serial diluted samples for a subset of HCV antibody reactive samples. Serial dilution of reactive samples will provide further insights into the potential difference of sensitivity in samples collected on DBS versus plasma.

Results of this trial will also support the update of the regulatory claims to include DBS as an alternative sample type.

DETAILED DESCRIPTION:
Access to Hepatitis C virus (HCV) screening in resource-limited settings should be enabled not only through the provision of point-of-care screening tests, but also through the possibility of collecting samples in decentralized settings One possible way of decentralizing sample collection is collecting dried blood spot (DBS) specimens, which can be easily transported to testing laboratories, not requiring any cold chain or complex sample transportation. DBS serology screening is complementary to established point-point-of care screening with rapid diagnostic tests, both methodologies being somewhat less cost-effective and less sensitive compared to lab-based methods but suitable for settings without sophisticated infrastructure.

To date, no HCV antibody serology test is formally evaluated for the use with DBS, however several studies on off-label use of DBS in serology screening assays, suggests that this sample type can serve as an alternative to plasma and serum. Fujirebio's enzyme immunoassay (EIA) INNOTEST® HCV Ab IV is CE marked and has received pre-qualification by the World Health Organization (WHO) for the use with venous plasma and serum, which require special equipment for sample collection, sample preparation and temperature controlled transportation.

Available data on the performance of HCV antibody detection from DBS samples are insufficient to introduce their use in clinical practice. Fujirebio is one of the few manufacturers who have an EIA test pre-qualified by the WHO for the use with plasma and serum to detect anti-HCV antibodies. A prospective diagnostic accuracy trial of the Fujirebio INNOTEST® HCV Ab IV assay in fWB and vWB collected on DBS, using EDTA plasma results obtained with the Fujirebio INNOTEST® HCV Ab IV assay as reference standard is needed to understand the relationship between results generated in plasma and WB samples collected on DBS. Furthermore, the data generated can be used by Fujirebio to update their regulatory claims and include DBS as an alternative sample type.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Provision of written informed consent
* Routine RDT reactive or non-reactive and recruitment target not yet met
* No history of HCV treatment

Exclusion Criteria:

* Unwilling to provide required volume of fingerstick blood and venous whole blood
* Participants already enrolled in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of fingerstick whole blood DBS | 4 months
  Point estimates of sensitivity and specificity (with 95% confidence intervals) of the Fujirebio INNOTEST® HCV Ab IV assay in fWB collected on DBS, using EDTA plasma results obtained with the Fujirebio INNOTEST® HCV Ab IV assay as reference standard
Sensitivity and specificity of venous whole blood DBS | 4 months
  Point estimates of sensitivity and specificity (with 95% confidence intervals) of the Fujirebio INNOTEST® HCV Ab IV assay in vWB collected on DBS, using EDTA plasma results obtained with the Fujirebio INNOTEST® HCV Ab IV assay as reference standard

SECONDARY OUTCOMES:
Degree of agreement of undiluted samples fWB and vWB | 4 months
  Point estimates of Cohen's Kappa Coefficient (ĸ) and negative, positive and overall rate of agreement of all undiluted samples for the Fujirebio INNOTEST® HCV Ab IV assay between fWB and vWB collected on DBS.
Degree of agreement of undiluted samples vWB and plasma | 4 months
  Point estimates of Cohen's Kappa Coefficient (ĸ) and negative, positive and overall rate of agreement of all undiluted samples for the Fujirebio INNOTEST® HCV Ab IV assay between vWB collected on DBS and plasma.
Degree of agreement of undiluted samples fWB and plasma | 4 months
  Point estimates of Cohen's Kappa Coefficient (ĸ) and negative, positive and overall rate of agreement of all undiluted samples for the Fujirebio INNOTEST® HCV Ab IV assay between fWB collected on DBS and plasma.
Degree of agreement of serial diluted samples fWB and vWB | 4 months
  Point estimates of Cohen's Kappa Coefficient (ĸ) and negative, positive and overall rate of agreement of serial-diluted HCV Ab positive samples for the Fujirebio INNOTEST® HCV Ab IV assay between fWB and vWB collected on DBS.
Degree of agreement of serial diluted samples vWB and plasma | 4 months
  Point estimates of Cohen's Kappa Coefficient (ĸ) and negative, positive and overall rate of agreement of serial-diluted HCV Ab positive samples for the Fujirebio INNOTEST® HCV Ab IV assay between vWB collected on DBS and plasma.
Degree of agreement of serial diluted samples fWB and plasma | 4 months
  Point estimates of Cohen's Kappa Coefficient (ĸ) and negative, positive and overall rate of agreement of serial-diluted HCV Ab positive samples for the Fujirebio INNOTEST® HCV Ab IV assay between fWB collected on DBS and plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Vasylyev, MD, Principal Investigator — Medical Centre Astar
Locations (2):
- Ukraine (2):
  - Astar Medical Centre, Lviv
  - Lviv Regional Public Health Centre, Lviv

IPD SHARING:
Plan to Share IPD: No